CLINICAL TRIAL: NCT02106533
Title: Effect of Aerobic Exercise Training on Ventilatory Efficiency in Patients With Coronary Artery Disease
Brief Title: Aerobic Exercise on Ventilatory Efficiency in CAD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital TotalCor (Other)
Responsible Party: Principal Investigator, Danilo Marcelo Leite do Prado, PHD, Hospital TotalCor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53/2010
Record Dates: First submitted 2014-03-27; First posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Coronary Artery Disease; Exercise Addiction; Complication, Cardio-respiratory
Keywords: Coronary artery disease; Exercise; Ventilatory efficiency
MeSH Terms: conditions — Coronary Artery Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 peak VO2 <17.5 ml/kg/min (Experimental): The exercise training program was comprised of three 60-minute exercise sessions per week over a 3-month period. Each exercise session consisted of a 5 minute warm up, 30-50 minutes of aerobic exercise performed on a treadmill and 5 minutes of cool-down exercises. Aerobic exercise intensity was set at the corresponding heart rate between the VAT and RCP.
  Interventions: Other: Aerobic exercise training
- Group 2 peak VO2 > 17.5 < 24.5 ml/kg/min (Experimental): The exercise training program was comprised of three 60-minute exercise sessions per week over a 3-month period. Each exercise session consisted of a 5 minute warm up, 30-50 minutes of aerobic exercise performed on a treadmill and 5 minutes of cool-down exercises. Aerobic exercise intensity was set at the corresponding heart rate between the VAT and RCP. All patients were able to achieve the set aerobic training intensity.
  Interventions: Other: Aerobic exercise training
- Group 3 peak VO2 > 24.5 ml/kg/min (Experimental): The exercise training program was comprised of three 60-minute exercise sessions per week over a 3-month period. Each exercise session consisted of a 5 minute warm up, 30-50 minutes of aerobic exercise performed on a treadmill . Aerobic exercise intensity was set at the corresponding heart rate between the VAT and RCP. All patients were able to achieve the set aerobic training intensity.
  Interventions: Other: Aerobic exercise training

INTERVENTIONS:
Other: Aerobic exercise training — The exercise training program was comprised of three 60-minute exercise sessions per week over a 3-month period. Each exercise session consisted of a 5 minute warm up, 30-50 minutes of aerobic exercise performed on a treadmill and 5 minutes of cool-down exercises. Aerobic exercise intensity was set at the corresponding heart rate between the VAT and RCP. All patients were able to achieve the set aerobic training intensity.

SUMMARY:
The purpose of the present study was to test the hypothesis that patients with coronary artery disease with lower aerobic fitness exhibit greater responsiveness on improving ventilatory efficiency after aerobic exercise training.

DETAILED DESCRIPTION:
Measurements of ventilatory efficiency during cardiorespiratory exercise testing typically expressed as the minute ventilation/ carbon dioxide production ratio have been validated to be useful in assessing the presence and severity of both heart and lung diseases. In this context, previous studies have showed ventilatory inefficiency in patients with coronary artery disease suggests abnormalities in the distribution of ventilation and perfusion in the lungs. In addition, a growing body of studies has demonstrated that lower ventilatory efficiency during exercise is considered an important predictor of risk mortality, hospitalization, and other outcomes than peak VO2.

ELIGIBILITY:
Inclusion Criteria:

* was stable coronary artery disease diagnosed by coronary angiography

Exclusion Criteria:

* unstable angina pectoris,
* complex ventricular arrhythmias,
* pulmonary congestion and
* orthopaedic or neurological limitations to exercise

Ages: 48 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Ventilatory efficiency in patients with coronary artery disease | up to 3 months of the interventions
  Measurements of ventilatory efficiency during cardiopulmonary exercise testing typically expressed as the minute ventilation/ carbon dioxide production ratio have been validated to be useful in assessing the presence and severity of both heart and lung diseases. In this context, previous studies have showed ventilatory inefficiency in patients with coronary artery disease suggests abnormalities in the distribution of ventilation and perfusion in the lungs.

CONTACTS AND LOCATIONS:
Overall Officials: Danilo ML Prado, PHD, Principal Investigator — Hospital TotalCor

REFERENCES:
- [Derived] Prado DM, Rocco EA, Silva AG, Silva PF, Lazzari JM, Assumpcao GL, Thies SB, Suzaki CY, Puig RS, Furlan V. The influence of aerobic fitness status on ventilatory efficiency in patients with coronary artery disease. Clinics (Sao Paulo). 2015 Jan;70(1):46-51. doi: 10.6061/clinics/2015(01)09. PMID 25672429